CLINICAL TRIAL: NCT05420597
Title: Induction Chemotherapy and Toripalimab Followed by Radiotherapy in Unresectable Laryngeal/Hypopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiayun He, MD, M.D., Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INSIGHT-2
Record Dates: First submitted 2022-06-12; First posted 2022-06-15 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Laryngeal Cancer; Hypopharyngeal Cancer
Keywords: Induction chemotherapy; Immunotherapy; Toripalimab; Radiotherapy
MeSH Terms: conditions — Laryngeal Neoplasms; Hypopharyngeal Neoplasms | interventions — toripalimab

STUDY DESIGN:
Intervention Model Description: Induction chemotherapy with toripalimab, followed by cisplatin-based concurrent chemoradiation. At 3-6 weeks post-radiation, maintenance toripalimab was administered for 8 cycles.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Induction chemotherapy and Toripalimab (Experimental): Induction chemotherapy TP regimen combined with Toripalimab, followed by cisplatin-based concurrent chemoradiation.
  Interventions: Drug: Toripalimab

INTERVENTIONS:
Drug: Toripalimab — Induction chemotherapy TP regimen combined with Toripalimab for 3 cycles: Toripalimab 240mg d1, Paclitaxel 175mg/m2 d2，Cisplatin 25mg/m2 d2-4 q3w. Then a total dose of 70Gy in 35 fractions was administered, with concurrently weekly cisplatin (30mg/m2 qw).
  At 3-6 weeks post-radiotherapy, maintenance Toripalimab was administered for 8 cycles (240mg d1 q3w, in total 8 cycles).
  Other Names: JS001

SUMMARY:
The aim of this study is to define whether combination of induction chemotherapy and PD-1 inhibitor (Toripalimab) followed by radiotherapy improve progression-free survival, for patients with unresectable laryngeal/hypopharyngeal carcinoma.

DETAILED DESCRIPTION:
Historically, induction chemotherapy has been shown to increase laryngeal-preservation rate, improve disease-free survival and reduce the risk of distant metastasis. However, the prognosis of locally advanced laryngeal/ hypopharyngeal carcinoma remains poor. Recently, phase I-II clinical studies demonstrated excellent pathological response of induction PD-1 inhibitor with/without chemotherapy for locally advanced head and neck cancer. The aim of this study is to define whether combination of induction chemotherapy and PD-1 inhibitor (Toripalimab) followed by radiotherapy improve progression-free survival, for patients with unresectable laryngeal/hypopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed, unresectable locally advanced laryngeal/hypopharyngeal squamous cell carcinoma due to extensively local invasion or medical comorbidities (T3-4b, N0-N3, M0);
* Age between 18-75 years;
* Signed inform consent;
* Had at least one measurable lesion according to RECIST 1.1 criteria
* Anticipated overall survival more than 3 months;
* Satisfactory performance status: ECOG (Eastern Cooperative Oncology Group) scale 0-1;
* Normal organ function and bone marrow function;
* HBV DNA<500 IU/mL（or 2500 copies/mL）and HCV RNA negative ;
* Male and no pregnant female, able to adapt birth control methods during treatment.

Exclusion Criteria:

* Hypersensitivity to Toripalimab, Paclitaxel or Cisplatin;
* Suffered from malignant tumors, except cervical carcinoma in situ, papillary thyroid carcinoma, or skin cancer (non- melanoma) within five years;
* Severe, uncontrolled heart disease;
* Receive vaccine or live vaccine within 28 days prior to signing the informed consent;
* Equivalent dose more than prednisone 10mg/d or other immunosuppressive treatments within 28 days prior to signing the informed consent;
* Surgery or trauma within 28 days prior to signing the informed consent;
* Received other immune checkpoint inhibitors previously;
* Severe, uncontrolled infections within 28 days of prior to signing the informed consent;
* Active, known or suspected autoimmune disease; Type I Diabetes, hypothyroidism those only need hormone replacement therapy, vitiligo or inactive asthma who don't need systemic therapy can recruit;
* History of interstitial lung disease;
* HIV positive;
* Hepatitis B surface antigen (HBsAg) positive and HBV-DNA ≥500IU/ml, or 2500cps/ml; Positive HCV RNA;
* Other diseases which may influence the safety or compliance of the clinical trial, such as mental illness, or their family and society factors;
* Women of child-bearing potential who are pregnant or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2021-04-07 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 2 year
  From the rate of enrollment to first progression

SECONDARY OUTCOMES:
Overall response rate of induction chemotherapy | up to 3 month
  Overall response rate of induction chemotherapy, evaluated by MR/CT imaging per RECIST 1.1
Locoregional recurrence-free survival | 2 year
  From the rate of enrollment to first locoregional relapse
Distant metastasis-free survival | 2 year
  From the rate of enrollment to first distant metastasis
Overall survival | 2 year
  From the rate of enrollment to death
Laryngeal Preservation Rate | 2 year
  The incidence of those with partial/whole preservation of anatomic larynx, without evidence of local recurrence
Adverse Effect | up to 2 year
  Adverse Effect, evaluated by CTCAE 4.0.03

CONTACTS AND LOCATIONS:
Overall Officials: Xiayun He, M.D., Principal Investigator — Fudan University; Yu Wang, M.D., Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No